CLINICAL TRIAL: NCT06960291
Title: Sustainable Implementation of the EXCEL Exercise Oncology Program Across Canada
Acronym: EXCEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other); Dalhousie University (Other); Nova Scotia Health Authority (Other); University of Toronto (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); University of British Columbia (Other); Memorial University of Newfoundland (Other); University of Prince Edward Island (Other); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-25-0029
Record Dates: First submitted 2025-04-04; First posted 2025-05-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Prostate Cancers; Breast Cancers; Colon Cancer; Lung Cancers
Keywords: Exercise oncology; Exercise; Physical activity; community program; online exercise; cancer survivor; individual living with and beyond cancer; quality of life
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Hybrid effectiveness-implementation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All participants will be involved in group exercise classes, twice a week for 8-12 weeks.
  Interventions: Behavioral: Group Exercise Classes

INTERVENTIONS:
Behavioral: Group Exercise Classes — Participants will take part in a combination of aerobic, resistance, balance, and flexibility exercises delivered in a circuit-type class setting, twice weekly for a 8-12-week period (duration of intervention depends on scheduling logistics for the coordinating hubs and their spokes sites). The exercise sessions will be conducted in groups with a ratio of up to 15 participants per instructor. The program follows exercise progression principles (i.e., frequency, intensity, time, type, overload and progression) over the 8-12-weeks, with tailoring of any exercise to meet individual participant needs as required, in order to promote fitness and wellness benefits.

SUMMARY:
EXCEL will provide online and, where feasible, in-person exercise programs to individuals living with and beyond cancer (ILWBC). Research has shown that targeted programs that include tailored exercise prescriptions are more successful in helping individuals with chronic disease to incorporate physical activity and exercise into their daily routines. While ILWBC are advised by healthcare professionals (HCPs) to engage in exercise, there is a lack of cancer-specific exercise programs and cancer-trained exercise specialists in Canada, outside of the research setting. Considering the negative impact cancer and its treatments have on fitness and physical activity levels, community-based efforts towards improving access, uptake and maintenance of exercise programming are needed.

This study will evaluate the benefits of a community-based or online EXCEL exercise program for people living with and beyond cancer across Canada, using a streamlined intake process compared to the original EXCEL Study (HREBA.CC-20-0098, NCT04478851). This 8 to 12-week program (intervention) will be delivered in-person or over virtual platform. It includes twice weekly supervised exercise classes.

DETAILED DESCRIPTION:
Over the past 4.5 years, the EXCEL Study (HREBA.CC-20-0098, NCT04478851) has been implemented across Canada and has recruited over 1500 individuals living with and beyond cancer. This updated study will streamline the program to essential baseline screening and testing (for safe and effective program delivery), simplify outcome assessments (for participants to see changes and for program evaluation), and increase the reach to include more urban centres to encourage more healthcare provider (HCP) buy-in with a simplified referral process (i.e. no patient screening required from HCPs to determine eligibility, based on location). This updated program is based off of the Alberta Cancer Exercise (ACE) Program (HREBA.CC-24-0252). Thus, we are modifying the original EXCEL ethics to will reduce the participant burden with less patient-reported-outcomes and fewer follow-ups, which will allow more focus on program implementation, evaluation, and sustainability. Continued effort and training to establish the clinic-to-community model will be enhanced with stronger relationships and referrals from the cancer care system and the HCPs, which will continue to work towards a 'patient-centered care approach'.

ELIGIBILITY:
Inclusion Criteria:

* have or had a diagnosis of cancer;
* be 18 years or older;
* be able to participate in low-intensity levels of activity, at minimum;
* be pretreatment, or receiving active cancer treatment (i.e., surgery, systemic therapy and radiation therapy), have received cancer treatment within the past 3 years, or if beyond 3 years since treatment completion, have a referral from their healthcare team indicating they have side effects from cancer treatment or the cancer itself, that could be improved or managed with exercise;
* be able to provide informed written consent in English or French

Exclusion Criteria:

* does not or did not have a cancer diagnosis
* is under the age of 18
* is unable to participate in mild exercise, at minimum
* is not pretreatment, or receiving active cancer treatment (i.e., surgery, systemic therapy and radiation therapy), has not received cancer treatment within the past 3 years, or if beyond 3 years since treatment completion, doesn't have side effects from cancer treatment or the cancer itself, that could be improved or managed with exercise
* unable to read/write in English
* for online programs, does not have internet or computer access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Level | Baseline to one year
  The Modified Godin Leisure Time Exercise Questionnaire is used to determine subjective levels of physical activity in each participant.

SECONDARY OUTCOMES:
Cancer related symptoms | Baseline to one year
  Change in Edmonton Symptom Assessment Scale - revised: cancer. Scale is from 0-10, where 0 means the symptom is absent and 10 means the worst possible severity of the symptom is being experienced.
Cost-effectiveness | Baseline to one year
  Change in EuroQual - 5Dimensions (EQ-5D) tool - first section is a questionnaire; last section uses a scale from 0-100, where 0 means the worst health imaginable and 100 means the best health imaginable.
Fatigue | Baseline to one year
  Change in Functional Assessment of Chronic Illness Therapy - Fatigue subscale - scale is from 0-4, where 0 means "not at all" and 4 means "very much".
Quality of life | Baseline to one year
  Single-item measure on quality of life - scale from 0 to 100, where 100 means the best Quality of Life imaginable and 0 means the worst Quality of Life imaginable.
Body Composition | Baseline to 12-weeks
  Change in body mass index (BMI)
Aerobic Capactiy | Baseline to 12-weeks
  Change in 6-minute walk test (m) or 2 minute step test (steps) results
Lower body strength | Baseline to 12-weeks
  Change in sit-to-stand (number of repetitions in 30 seconds)
Upper extremity flexibility | Baseline to 12-weeks
  Change in active shoulder flexion range of motion (degrees)
Balance | Baseline to 12-weeks
  Change in one legged stance test (seconds)
Exercise adherence | Duration of the intervention (8-12 week exercise program)
  Adherence to exercise programming (attendance at sessions)
Program implementation and evaluation | Baseline to one year
  RE-AIM: program reach, effectiveness, adoption, implementation and maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Culos-Reed, PhD, Principal Investigator — University of Calgary
Locations (5):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - University of Toronto, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
No plan at this time to share IPD outside of the research team.